CLINICAL TRIAL: NCT05542186
Title: Immediate Effects of Kinesio Taping on Pain and Postural Stability in Persons With Discogenic Low Back Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/11
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kinesiotaping (Experimental)
  Interventions: Procedure: Kinesiotaping

INTERVENTIONS:
Procedure: Kinesiotaping — Biomechanical correction for discogenic low back pain using kinesiotaping

SUMMARY:
Discogenic LBP is the leading cause of disability worldwide. Eventhough other types of Chronic LBP are more common, 63% of all patients reporting to tertiary care hospital with LBP are discogenic in nature. However, immediate effects of kinesio-taping on pain and postural stability in discogenic low back pain has not been well documented in existing literature. This study is focused on immediate effects of kinesiotaping on pain and postural stability in persons with discogenic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants in an age range of 20-65 years will be considered for this study.
* Participants with disc bulge, herniation or prolapse indicate by MRI.
* Positive straight leg raise (SLR) Positive centralization and peripheralization phenomenon.
* Participants with MRI findings conclusive of disc pathology will be included.

Exclusion Criteria:

-

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Pain Pressure Threshold | 1 day
  Pain Pressure Threshold will be measured using algometer before and after the treatment session. Higher score signifies positive outcome.
Back Pain | 1 day
  Pain will be measured using numeric pain rating scale before and after the treatment session. Higher score signifies negative outcome.
Postural Stability | 1 day
  Postural Stability will be measured using Biodex Balance System before and after the treatment session

CONTACTS AND LOCATIONS:
Overall Officials: Bisma Mazhar, MS, Principal Investigator — FUI; Muhammad Osama, PhD*, Study Chair — FUI
Locations (1):
- Foundation University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No